CLINICAL TRIAL: NCT05798494
Title: PRE-Pregnancy Weight Loss And the Reducing Effect on CHILDhood Overweight - Aarhus
Acronym: PREPARE CHILD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ulla Kampmann Opstrup (Other)
Collaborators: Per Ovesen, Professor Dept. of Obsteterics, Aarhus University Hospital (Unknown); Jens Meldgaard Bruun, Professor Steno Diabetes Center Aarhus, Aarhus University Hospital (Unknown); Sine Knorr, PhD Steno Diabetes Center Aarhus, Aarhus University Hospital (Unknown)
Responsible Party: Sponsor-Investigator, Ulla Kampmann Opstrup, Associate professor, Aarhus University Hospital
Organization: University of Aarhus (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Prepare Child AUH
Record Dates: First submitted 2023-02-21; First posted 2023-04-04 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Overweight and Obesity; Weight Loss; Pregnancy Related; Child Nutrition Sciences; Body Composition
Keywords: Overweight; Pregnancy; Weight loss; Diet, Reducing; Epigenetics; Healthy Lifestyle; DNA Methylation; Exercise; Offspring's neonatal fat mass; Pea Pod; Infant, Large for Gestational Age; Body Fat Distribution
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Motor Activity

STUDY DESIGN:
Intervention Model Description: 140 couples will be recruited and randomized to either intervention og control. Participants includes the mother, father and 1st and 2nd child, therefore the total number of participants will be 560.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention group will receive dietary counseling by a trained dietitian from 3 months post-partum of the 1st child until birth of the 2nd child. The mother will receive advice to provide a moderate caloric restriction (-500 to 1000 kcal/d) and attend physical activity sessions to attain a 10 % weight loss according to pre-pregnancy weight. If the father is also overweight or obese, he will receive the same advice.
  Interventions: Behavioral: Weight loss intervention
- Control (No Intervention): The control group will receive standard care and will not receive any dietary advice prior to pregnancy. During pregnancy control subjects will receive dietary advice according to standard care which means no counselling from a dietitian unless there are special needs (e.g., gestational diabetes), then they will receive counseling from a dietitian in accordance with standard care.

INTERVENTIONS:
Behavioral: Weight loss intervention — Subjects will receive dietary counseling by a dietitian from 3 months post-partum of the 1st child until birth of the 2nd child. The mother (and father if overweight, BMI ≥25 kg/m^2) will receive advice to provide a moderate caloric restriction (-500 to 1000 kcal/d) and power walk 2-4 times a week for a half an hour and attend physical activity sessions every 2nd week to attain a minimum weight loss of approximately 0,5-1,0 kg/week. The weight loss will last until a 10% weight loss (according to pre-pregnancy weight) has been achieved or until 1-year post-partum. If the subject has not achieved a weight loss of 10%, she or he will receive Very low-calorie diet (VLCD) until target weight loss is reached, though no longer than 8 weeks. After weight loss subjects will receive counseling to maintain weight loss and healthy weight gain during pregnancy until birth of the 2nd child.
  Arms: Intervention

SUMMARY:
The study is a single site parallel randomized controlled study. The study will be assessing the effect of a 10% pre-conceptional weight loss intervention vs a control group among healthy couples where the prospective mother is pregnant and overweight or obese (BMI 27-44.9 kg/m^2). The couples in intervention group will receive dietitian counseling and participate in physical activity sessions to attain the 10% weight loss. The overall objective is to test whether a comprehensive pre-conceptional parental weight loss intervention effectively reduces the risk of offspring overweight, and adiposity and its complications compared to a control group.

DETAILED DESCRIPTION:
The study is a single site parallel randomized controlled study. The study will be assessing the effect of a pre-conceptional weight loss intervention vs a control group among healthy couples where the prospective mother is pregnant (recruited at gestational age 18-36), overweight or obese (BMI 27-44.9 kg/m^2), between 18-38 years and planning an additional pregnancy within the following 3 years.

The investigators will recruit a total of 140 healthy pregnant couples who will be randomized 1:1 to either intervention or control, stratified according to maternal pre-pregnancy BMI and previous or present diagnosis of gestational diabetes.

The couples in intervention group will receive dietary counseling by a dietitian from 3 months post-partum of the 1st child until birth of the 2nd child. The goal is to achieve a healthy lifestyle and a moderate weight loss of 10% according to pre-pregnancy weight during the first year. Hereafter, the couples will be guided in weight maintenance until pregnancy of the second child. During pregnancy the goal is to achieve a healthy weight gain. Couples in intervention group will also participate in physical activity sessions every 2nd week and advised to walk with moderate intensity at least 2-4 times a week for at least half an hour.

The overall objective is to test whether a comprehensive pre-conceptional parental weight loss intervention effectively reduces the risk of offspring overweight, and adiposity and its complications compared to a control group. The 1st baby born before intervention is started will be the "index child" and the metabolic and anthropometric parameters of the 1st child will be compared to parameters of the second child to assess the effect of the parent's healthy lifestyle between the two pregnancies.

The investigators hypothesize that parental weight loss intervention, initiated before conception, will facilitate lower parental insulin resistance, inflammation, body weight and adiposity, incretin responses and energy expenditure compared to usual care. For the offspring the investigators hypothesize that the intervention will reduce adverse pregnancy outcomes with a short-term reduction in the risk of being born large for gestational age with excessive fat mass and a long-term reduction in the risk of developing overweight or obesity as a consequence of both social (family approach) and biological (epigenetic modifications) pathways.

ELIGIBILITY:
Maternal inclusion Criteria:

* Maternal pre-pregnancy BMI 27.0-44.9 kg/m^2
* Maternal age range 18-38 years
* Connected to Aarhus University Hospital as place of birth
* Pregnant

Paternal Inclusion Criteria:

* Paternal pre-pregnancy BMI 18.5-44.9 kg/m^2
* Paternal age range 18-55 years

Parental Inclusion Criteria:

* Couples (male and female)
* Planning pregnancy within 3 years
* Provided voluntary informed consent
* Danish or English speaking
* Intention to permit the planned offspring to participate in the follow-up study
* Able to store biological samples from the offspring at home in the freezer in a box given by the study personnel

Parental Exclusion Criteria:

* Diabetes mellitus (Type 1 or 2)
* Previous or present eating disorder
* Allergy towards ingredients in the very low calorie diet products
* Severe heart, liver or kidney disease
* Conception by in vitro fertilization
* Any medical condition or concomitant medication as judged by the medical responsible
* Adherence to vegan diets or other diets interfering with the dietary guidelines in the study
* Participation in other clinical trial that can affect the results of the current study
* Engagement in elite sports or similar strenuous exercise ≥5 h/week at inclusion
* Blood donation or transfusion within the past month before screening
* Blood donation during the study
* Inability or unwillingness to follow the study protocol and instructions given by the study personnel

A detailed description of the exclusion criteria is given below:

Medical conditions as known by the participant:

* Diabetes mellitus (type 1 and 2)
* History or diagnosis of eating disorder (e.g. restrained eating, disinhibition, emotional eating)
* Any significant medical condition as assessed by the investigator (e.g. dysregulated thyroid disease or reproductive diseases)
* Any significant psychiatric disorder (i.e. schizophrenia, bipolar disease or depression) as assessed by the investigator
* Severe chronic heart, liver and kidney disease
* Polycystic ovary syndrome with irregular cycle

Medication:

* Current use of medication or use within the previous three months with a potential to affect body weight or pregnancy as judged by the investigator (e.g. systemic corticoids)

Personal/other:

* Severe food allergies, food intolerances or dislike expected to interfere with the study, including allergy towards ingredients in the VLCD products
* Engagement in elite sports or similar strenuous exercise ≥5 h/week
* Blood donation or transfusion within the past month before screening
* Planned blood donation for other purpose than this study during participation
* Alcohol abuse, as judged by the investigator, within the previous 12 months
* Drug abuse, as judged by the investigator, within the previous 12 months
* Psychological or behavioral problems which, in the judgement of the investigator, would lead to difficulty in complying with the study protocol
* Participation in other clinical trials within the past three months or intention to do so during the study, which are judged by the investigator to affect the present study
* Unable to consume the interventional product for religious reasons, swallowing disorders, other physiological reasons or any other reasons for not being able to follow the recommended diet
* Inability or unwillingness to give written informed consent or communicate with study personnel
* Inability or unwillingness to follow the study protocol and instructions given by the study personnel
* Illiteracy or inadequate understanding of Danish or English language.
* Any other condition that judged by the investigator may interfere with the adherence to the study protocol

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-04-11 (Estimated); Study Completion 2028-04-11 (Estimated)

PRIMARY OUTCOMES:
Neonatal fat mass | Collected within the first week of birth (strived <48 hours)
  Offspring's neonatal fat mass (grams) assessed by air displacement plethysmography (Pea POD)
Difference in epigenetic changes in child 1 and 2 | Assessed at birth
  Cord blood from offspring will be collected at birth and stored at -80 °C until use. At the Department of Molecular Medicine AUH genomic DNA will be extracted from peripheral blood using standard methods e.g., QIAmp® Mini Kit (Qiagen, Germany). 1 μg of genomic DNA will be bisulfide converted using Illumina iScan (platform). The methylation level will be measured using Infinium MethylationEPIC DNA Analysis BeadChip (Array type) at Eurofins Genomics AS (Denmark) or similar methods.
  The stated required sample size (140 couples) is calculated based on the neonatal fat mass. As no other studies have performed methylation analysis using WGBS in similar cohorts, precise power calculations on epigenetic changes are impractical. However, since the EPICOM study found differentially methylated regions in only 20 cases and 20 controls using Illumina's 450K methylation assay, the power to elucidate epigenetic changes is considered sufficient in the planned study.

SECONDARY OUTCOMES:
Obstetrics outcome - length of gestational age | Assessed at birth of both offsprings
  Length of gestational age
Obstetric - medication use | Collected from initiation of labor until completed birth of both offsprings
  Medication use during labor
Obstetric - delivery mode | Collected at birth of both offsprings
  Delivery mode (rupture of membranes or premature contractions, vaginal, cesarean section, instrumental delivery, miscarriage and stillbirth).
Obstetric - pregnancy complications | Collected at gestational age (GA) 34-36 and after birth of both offsprings
  Pregnancy complications e.g. miscarriage, abortion (induced and indication for abortion), hydramnios, gestational hypertension, preeclampsia, need for maternal corticosteroid treatment for fetal lung maturation, urinary tract infection) will be collected from medical record.
Obstetric - Neonatal unit admissions | Collected at birth and until 12 months after birth of both offsprings
  Neonatal unit admissions
Obstetric - obstetrics complications | Collected at birth of both offsprings
  Obstetrics complications (e.g. preterm prelabour rupture of the membranes, shoulder dystocia, birth trauma (perinatal rupture), postpartum hemorrhage, maternal infections, maternal hospitalization).
Obstetrics - birth defects/abnormalities | Collected at birth of both offsprings
  Birth defects/abnormalities
Neonatal morbidities | Collected at birth of both offsprings
  Neonatal morbidity (e.g. major congenital malformations (ICD10 Q00-Q99 or requiring medical or surgical treatment), birth injury, respiratory distress, transient tachypnoea, neonatal hypoglycemia, systemic infections, admission to neonatal intensive care unit, number of admission days, hyperbilirubinemia), deaths.
Fetal and offspring growth - body weight | Collected from medical record during pregnancy, measured in gestational age (GA) GA34-GA36 via ultrasound in both pregnancies, at birth and 3, 12 and 18 months after birth of both offsprings
  Fetal body weight will be measured with ultrasound during pregnancy and offspring body weight will be measured using an electronic scale.
Fetal and offspring growth - length | Collected from medical record during pregnancy, measured in GA34-GA36 via ultrasound in both pregnancies, and measured at birth and 3, 12 and 18 months after birth of both offsprings
  Fetal length will be measured with ultrasound during pregnancy and offspring length will be measured using an infantometer as appropriate for measuring infant, baby and toddler length.
Fetal and offspring growth - abdominal circumference | Collected from medical record during pregnancy, measured in GA34-GA36 via ultrasound in both pregnancies, and measured at birth and 3, 12 and 18 months after birth of both offsprings
  Abdominal circumference will be measured with ultrasound during pregnancy and offspring abdominal circumference will be measured three times to the nearest 0.1 cm using a stretch-resistant measuring tape
Fetal and offspring growth - crown circumference | Collected from medical record during pregnancy, measured in GA34-GA36 via ultrasound in both pregnancies
  Crown circumference will be measured with ultrasound during pregnancy
Fetal and offspring growth - femur length | Collected from medical record during pregnancy, measured in GA34-GA36 via ultrasound in both pregnancies,
  Femur length will be measured with ultrasound during pregnancy
Fetal growth - fractional limb volume | Collected from medical record during pregnancy, measured in GA34-GA36 via ultrasound in both pregnancies,
  Fractional limb volume will be measured with ultrasound during pregnancy
Offspring growth - BMI z-score | Collected at birth and 3, 12 and 18 months after birth of both offsprings
  Offspring body mass index (BMI) z-score (BMI adjusted for age and sex).
Offspring growth - weight for gestational age | Collected at birth and 3, 12 and 18 months after birth of both offsprings
  Weight for gestational age. Measured as percent of normal weight related to gestational age.
Offspring growth - large for gestational age | Collected at birth of both offsprings
  Large for gestational age. Prevalence of infants being large for gestational age (LGA).
Offspring growth - small for gestational age | Collected at birth of both offsprings
  Small for gestational age. Prevalence of offspring being small for gestational age (SGA).
Offspring growth - apgar score | Collected at birth of offspring of both offsprings
  Apgar score (0-10). The higher the score, the better health condition of the offspring)
Offspring growth | Collected at birth and 3, 12 and 18 months after birth of offspring.
  Offspring circumference (thigh and upper arm) and skinfold (triceps, subscapularis and suprailiac). Circumferences will be measured to the nearest 0.1 cm using a stretch-resistant measuring tape and skinfolds are measured to the nearest 0.02 cm using a caliper to lightly pinch the skin and the underlying fat.
Offspring growth - body composition by the POD system | Collected within the first week of birth and 3 months post partum in both offsprings
  Offspring fat free mass (g) and fat mass (g) will be assessed by air displacement plethysmography using the POD system (Pea POD for 1-8kg)
Offspring blood pressure | Collected 12 and 18 months after birth of both offsprings
  Offspring blood pressure (diastolic and systolic blood pressure) will be measured three times after 10 minutes rest using an automated device placed on the arm and in direct contact with the skin.
Offspring heart rate | Collected 12 and 18 months after birth of both offsprings
  Offspring heart rate will be measured three times after 10 minutes rest using an automated device placed on the arm and in direct contact with the skin.
Offspring growth - self-reported body weight | 18 months after birth the study staff will make an annual follow-up phone call to the parents to collect information about the offspring's self-reported body weight until the offspring is 18 of age
  Self-reported body weight
Offspring growth - self-reported height | 18 months after birth the study staff will make an annual follow-up phone call to the parents to collect information about the offspring's self-reported body weight until the offspring is 18 of age
  Self-reported height
Adult weight | Intervention: each visit throughout study (GA34-36 of 1st child to 18mo. after birth of 2nd child). Control: In GA34-36 in both pregnancies, at study visits (3, 12 and 24mo. pp) and follow up visits (3, 12 and 18 months pp of 2nd child)
  Adult body weight is measured to the nearest 0.1 kg using a calibrated scale
Adult Height | Collected in GA34-GA36 in index pregnancy
  Adult height will be measured to the nearest 0.5 cm using a wall-mounted stadiometer.
Adult BMI | Collected in GA34-36 in 1st pregnancy, study visits 3, 12 and 24mo. pp after 1st child, GA34-36 in 2nd pregnancy and at follow up vist (3, 12 and 18mo. pp of 2nd child).
  Calculated as weight (kg)/height(m)^2
Adult anthropometric | Intervention: each visit throughout study (GA34-36 of 1st child to 18mo. after birth of 2nd child). Control: In GA34-36 in both pregnancies, at study visits (3, 12 and 24mo. pp) and follow up visits (3, 12 and 18 months pp of 2nd child)
  Waist- and hip circumference will be measured to the nearest 0.1 cm. During pregnancy and at birth the waist of the female will not be measured.
Adult blood pressure | Collected at GA34-36 in 1st pregnancy, study visits 3, 12 and 24 months pp. of 1st child, GA34-36 in 2nd pregnancy and 3 months pp after 2nd child
  Blood pressure (diastolic and systolic blood pressure) will be measured three times with two minutes apart in right arm after 15 minutes rest using a validated automatic device. The reading is recorded to the nearest 1 mmHg.
Adult heart rate | Collected at GA34-36 in 1st pregnancy, study visits 3, 12 and 24 months pp. of 1st child, GA34-36 in 2nd pregnancy and 3 months pp after 2nd child
  Heart rate will be measured three times with two minutes apart in right arm after 5-10 minutes rest using a validated automatic device. The reading is recorded to the nearest 1 beats/minute for heart rate
Adult resting metabolic rate | Collected at study visit 3, 12, and 24 months pp after 1st child.
  Resting metabolic rate (calories/24-h) will be measured by indirect calorimetry using a ventilated hood system. Participants will lie in the supine position and rest for at least 30 min before measurements commence. The measurement will last for 20 min.
Adult resting respiratory quotient + substrate | Collected at study visit 3, 12, and 24 months pp after 1st child.
  Resting respiratory quotient (RQ), will be measured by indirect calorimetry using a ventilated hood system. Participants will lie in the supine position and rest for at least 30 min before measurements commence. The measurement will last for 20 min. Lipid, glucose and protein oxidation will be estimated.
Adult medication use | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st. child
  Use of medication will be collected throughout the study and for each medication the start date, stop date or continuing, form and indication will be noted in appropriate form.
Offspring medication use | Birth, after 3, 12, and 18 months after birth of both offsprings
  Use of medication will be collected throughout the study and for each medication the start date, stop date or continuing, form and indication will be noted in appropriate form.
Adult reproduction - Time to pregnancy | Registration of 2nd. pregnancy (up to tree years from birth of 1.st. child)
  Duration of time to conception defined from selfreported time point they started to try get pregnant to registration of pregnancy. The time of conception will be calculated from the ultrasound scan in week 12
Adult glucose metabolism (OGTT) | Performed at study visits 3, 12 and 24 months pp of 1st. child
  3-h oral glucose tolerance test (OGTT) will be performed at with 75g of glucose dissolved in 250 ml of water and added 1 gram of paracetamol. Blood will collected for measurements of blood glucose, hormones (insulin, C-Peptide, glucagon), paracetamol, glucagon-like-peptide-1 (GLP-1), Glucose insulinotropic polypeptide (GIP) and metabolites (FFA). Blood samples will be drawn at time 0, 15, 30, 45, 60, 90, 120 and 180 min
Adult Oral Glucose Tolerance Test (OGTT) during pregnancy (only female) | Collected in GA28 of 1st and 2nd pregnancy (performed after risk score at gestational age~20 and ~28 or only ~28)
  OGTT performed during pregnancy according to the screening guidelines for GDM will be obtained from the mother's medical journal in both pregnancies.
Placenta - weight (gram) | Collected at birth of both offsprings
  Placenta will be weighted after birth
VO2-max adult - cardiorespiratory fitness | Collected at study visit 3, 12 and 24 months pp after birth of 1st child
  The VO2-max test will be performed as an incremental exercise test on a bicycle ergometer.
Cardiac function offspring - Left ventricular and right ventricular morphology | Collected at birth and at 12 months follow up visit after birth of each child
  ECG and echocardiography will be performed according to standard imaging protocol. Assessment of Interventricular septal thickness diastole and valve- and chamber dimensions will be done.
Cardiac function offspring - left centricular ejection fraction | Collected at birth and at 12 months follow up visit after birth of each child
  ECG and echocardiography will be performed according to standard imaging protocol. Assessment of left ventricular ejection fraction will be done.
Cardiac function offspring - fractional shortening | Collected at birth and at 12 months follow up visit after birth of each child
  ECG and echocardiography will be performed according to standard imaging protocol. Assessment of fractional shortening will be done.
Cardiac function offspring - Systolic function, strain | Collected at birth and at 12 months follow up visit after birth of each child
  ECG and echocardiography will be performed according to standard imaging protocol. Assessment of strain will be done.
Cardiac function offspring - Systolic function, strain rate | Collected at birth and at 12 months follow up visit after birth of each child
  ECG and echocardiography will be performed according to standard imaging protocol. Assessment of strain rate will be done.
Cardiac function offspring - TAPSE and RV fractional area change | Collected at birth and at 12 months follow up visit after birth of each child
  ECG and echocardiography will be performed according to standard imaging protocol. Assessment of TAPSE and RV fractional area change will be done.
Cardiac function offspring - Diastolic function, left ventricular E/A-ratio | Collected at birth and at 12 months follow up visit after birth of each child
  ECG and echocardiography will be performed according to standard imaging protocol. Assessment of left ventricular E/A-ratio will be done.
Cardiac function offspring - Diastolic function, tissue velocities (E', A', S') | Collected at birth and at 12 months follow up visit after birth of each child
  ECG and echocardiography will be performed according to standard imaging protocol. Assessment of tissue velocities (E', A', S') will be done.
Cardiac function offspring - Diastolic function, strain | Collected at birth and at 12 months follow up visit after birth of each child
  ECG and echocardiography will be performed according to standard imaging protocol. Assessment of strain will be done.
Cardiac function offspring - Overall cardiac function | Collected at birth and at 12 months follow up visit after birth of each child
  ECG and echocardiography will be performed according to standard imaging protocol. Assessment of Myocardial performance index (MPI) and cardiac torsion will be done.
Cardiac function offspring - Pulmonary artery acceleration time | Collected at birth and at 12 months follow up visit after birth of each child
  ECG and echocardiography will be performed according to standard imaging protocol. Assessment of Pulmonary artery acceleration time will be done.
Cardiac function offspring - Pulmonary artery pressure | Collected at birth and at 12 months follow up visit after birth of each child
  ECG and echocardiography will be performed according to standard imaging protocol. Assessment of Pulmonary artery pressure will be done.
Cardiac function offspring - Persistent ductus arteriosus (PDA) | Collected at birth and at 12 months follow up visit after birth of each child
  ECG and echocardiography will be performed according to standard imaging protocol. Assessment of PDA open or closed and PDA shunt will be done.
Cord blood - Telomore length | Collected at birth of both offsprings
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for Telomore length.
Cord blood - pH | Collected at birth
  Cord blood will be drawn immediately after birth. pH will be assessed.
Cord blood - Epigenetics | Collected at birth of both offsprings
  Epigenetics analyses from whole blood. Will be analysed for methylation changes. metabolomics and exosome.
Adult body composition by DEXA scan | Collected at study visits 3, 12 and 24 months pp. of 1st child
  Lean mass (g), fat mass (g), abdominal fat (g), visceral fat (g) assessed by a Dual-energy X-ray absorptiometry (DEXA) -scan .
Adult bone markers by DEXA scan - bone mineral content | Collected at study visits 3, 12 and 24 months pp. of 1st child
  Bone mineral content (g) assessed by a Dual-energy X-ray absorptiometry-scan.
Adult bone markers by DEXA scan - bone area | Collected at study visits 3, 12 and 24 months pp. of 1st child
  Bone area (cm^2) assessed by a Dual-energy X-ray absorptiometry-scan.
Adult bone markers by DEXA scan - bone mineral density | Collected at study visits 3, 12 and 24 months pp. of 1st child
  Bone mineral density (g/cm^2) assessed by a Dual-energy X-ray absorptiometry-scan.
Adult blood sample - glucose | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for glucose
Adult blood sample - CD163 | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for CD163
Adult blood sample - HbA1c | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for markers of glucose metabolism HbA1c
Adult blood sample - Kreatinin | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for kreatinin
Adult blood sample - eGFR | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for kreatinin and GFR will be estimated
Adult blood sample - C-reaktivt protein (CRP) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for CRP
Adult blood sample - Alanintransaminase (ALAT) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for ALAT
Adult blood sample - Gamma-GT (GGT) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for GGT
Adult blood sample - Basisk fosfatase (BASP) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for BASP
Adult blood sample - Bilirubin | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for Bilirubin
Adult blood sample - Ferritin | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for Ferritin
Adult blood sample - Hemoglobin | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for Hemoglobin
Adult blood sample - Leukocytter | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for Leucocytter
Adult blood sample - platelets | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for platelets
Adult blood sample - Triglyceride | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for triglyceride
Adult blood sample - Cholesterol HDL | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for Cholesterol HDL
Adult blood sample - Cholesterol LDL | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for Cholesterol LDL
Adult blood sample - Total Cholesterol | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for Total Cholesterol
Adult blood sample - vitamin B12 | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for B12
Adult blood sample - vitamin D3 | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for vitamin D3
Adult blood sample - c-peptide | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for c-peptide
Adult blood sample - Insulin-like Growth Factor-1 (IGF-1) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for IGF-1
Adult blood sample - Insulin-like growth factor-binding protein-1 (IGFBP-1) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for IGFBP-1
Adult blood sample - Insulin-like growth factor-binding protein-3 (IGFBP-3) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for IGFBP-3
Adult blood sample - Fibroblast growth factor 21 (FGF-21) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for FGF-21
Adult blood sample - Leptin | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for Leptin
Adult blood sample - Adiponectin | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for Adiponectin
Adult blood sample - Ghrelin | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for Ghrelin
Adult blood sample - Growth Hormone (GH) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for GH
Adult blood sample - Free fatty Acids (FFA) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for FFA
Adult blood sample - Interleukin 6 (IL-6) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for IL-6
Adult blood sample - Interleukin 6 (IL-10) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for IL-10
Adult blood sample - Interleukin-1 alpha (IL-1 alpha) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for IL-1 alpha
Adult blood sample - Interferon gamma (IFN-γ) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for IFN-γ
Adult blood sample - Tumor Necrosis Factor alfa (TNF-α) | Collected at GA34-GA36 in 1st pregnancy, study visit 3, 12 and 24 months pp of 1st child, at GA34 in 2nd pregnancy and at follow visit 3 months pp after 2nd child
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for TNF-α
Adult female blood sample - Humant choriogonadotropin (hCG) | Collected at GA34-GA36 in both pregnancies
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will only be collected from the female participant during pregnancy and be analysed for hCG
Adult female blood sample - Progesterone | Collected at GA34-GA36 in both pregnancies
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will only be collected from the female participant during pregnancy and be analysed for Progesterone
Adult female blood sample - Proinsulin C-peptide | Collected at GA34-GA36 in both pregnancies
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will only be collected from the female participant during pregnancy and be analysed for Proinsulin C-peptide
Adult female blood sample - sex hormone binding globulin (SHBG) | Collected at GA34-GA36 in both pregnancies
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will only be collected from the female participant during pregnancy and be analysed for SHBG
Adult female blood sample - Prolactin | Collected at GA34-GA36 in both pregnancies
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will only be collected from the female participant during pregnancy and be analysed for Prolactin
Adult blood sample -Cortisol | Collected at GA34-GA36 in both pregnancies
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will be analysed for Cortisol
Adult female blood sample -Estradiol | Collected at GA34-GA36 in both pregnancies
  All blood samples will be collected by venous puncture in the antecubital vein after an overnight fast from at least 10 pm the night before. Samples will only be collected from the female participant during pregnancy and be analysed for Estradiol
Offspring blood sample - glucose | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for glucose
Offspring blood sample - c-peptide | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for c-peptide
Offspring blood sample - insulin | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for Insulin
Offspring blood sample - IGF-1 | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for IGF-1
Offspring blood sample - IGFBP-3 | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for IGFBP-3
Offspring blood sample - IGFBP-1 | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for IGFBP-1
Offspring blood sample - CD163 | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for CD163
Offspring blood sample - Ferritin | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for Ferritin
Offspring blood sample - HgbA1c | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for HgbA1c
Offspring blood sample - Hgb | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for Hgb
Offspring blood sample - CRP | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for CRP
Offspring blood sample - Triglyceride | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for Triglyceride
Offspring blood sample - Cholesterol HDL | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for Cholesterol HDL
Offspring blood sample - Cholesterol LDL | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for Cholesterol LDL
Offspring blood sample - Total Cholesterol | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for Total Cholesterol
Offspring blood sample - FGF-21 | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for FGF-21
Offspring blood sample - Leptin | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for Leptin
Offspring blood sample - Adiponectin | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for Adiponectin
Offspring blood sample - FFA | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for FFA
Offspring blood sample - Growth Hormone (GH) | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for GH
Offspring blood sample - cTroponin I (cTnI) | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for cTnI
Offspring blood sample - BNP | Collected 12 months after birth in both offsprings
  A non-fasting venous blood will be drawn. Parents will be instructed that the offspring should not have eaten two hours prior to the assessment. Samples will be analysed for BNP
Cord blood - c-peptide | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for C-peptide
Cord blood -Insulin | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for Insulin
Cord blood -IGFBP-3 | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for IGFBP-3
Cord blood -IGFBP-1 | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for IGFBP-1
Cord blood -IGF-1 | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for IGF-1
Cord blood -Ferritin | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for Ferritin
Cord blood -cTnI | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for cTnI
Cord blood -BNP | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for BNP
Cord blood -CRP | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for CRP
Cord blood -CD163 | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for CD163
Cord blood -FGF21 | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for FGF21
Cord blood -Leptin | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for Leptin
Cord blood -Adiponectin | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for Adiponectin
Cord blood -FFA | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for FFA
Cord blood - Vitamin D3 | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for Vitamin D3
Cord blood - HbA1c | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for HbA1c
Cord blood - IL-6 | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for IL-6
Cord blood - IL-10 | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for IL-10
Cord blood - IL-1 alpha | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for IL-1 alpha
Cord blood -TNF- alpha | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for-TNF- alpha
Cord blood -IFN- gamma | Collected at birth of both offspring
  Cord blood will be drawn immediately after birth and analysed. Blood will be analyzed for IFN- gamma

OTHER OUTCOMES:
Offspring feces - Microbiome | Collected within the first week after birth (but should avoid to collect the first fecal excretion after birth (meconium)), at study visit 3 and 12 months after birth of each offspring
  Will be analysed for microbiome. Collected at birth by researcher and home by parents preferable <24 hours before the planned visit.
Offspring feces - Short chain fatty acids | Collected within the first week after birth (but should avoid to collect the first fecal excretion after birth (meconium)), at study visit 3 and 12 months after birth of each offspring
  Will be analysed for short chain fatty acids. Collected at birth by researcher and home by parents preferable <24 hours before the planned visit.
Offspring feces - Metabolomics | Collected within the first week after birth (but should avoid to collect the first fecal excretion after birth (meconium)), at study visit 3 and 12 months after birth of each offspring
  Will be analysed for metabolomics. Collected at birth by researcher and home by parents preferable <24 hours before the planned visit.
Offspring feces - Proteomics | Collected within the first week after birth (but should avoid to collect the first fecal excretion after birth (meconium)), at study visit 3 and 12 months after birth of each offspring
  Will be analysed for proteomics. Collected at birth by researcher and home by parents preferable <24 hours before the planned visit.
Offspring feces - pH | Collected within the first week after birth (but should avoid to collect the first fecal excretion after birth (meconium)), at study visit 3 and 12 months after birth of each offspring
  Will be assessed for pH. Collected at birth by researcher and home by parents preferable <24 hours before the planned visit.
Offspring feces - Inflammation markers | Collected within the first week after birth (but should avoid to collect the first fecal excretion after birth (meconium)), at study visit 3 and 12 months after birth of each offspring
  Will be analysed for inflammation markers. Collected at birth by researcher and home by parents preferable <24 hours before the planned visit.
Offspring feces - consistency | Collected within the first week after birth (but should avoid to collect the first fecal excretion after birth (meconium)), at study visit 3 and 12 months after birth of each offspring
  Whenever a fecal sample is collected stool consistency of the collected sample will be collected with a questionnaire.
Offspring feces - frequency | Collected within the first week after birth (but should avoid to collect the first fecal excretion after birth (meconium)), at study visit 3 and 12 months after birth of each offspring
  Whenever a fecal sample is collected an estimate of stool frequency during the last week will be collected with a questionnaire.
Offspring feces - gastrointestinal symptoms | Collected within the first week after birth (but should avoid to collect the first fecal excretion after birth (meconium)), at study visit 3 and 12 months after birth of each offspring
  Whenever a fecal sample is collected any gastrointestinal symptoms of the offspring during the last week will be collected with a questionnaire.
Offspring urine | Collected within the first week of birth and at 3 and 12 months follow up of each offspring
  Parents will be instructed to collect offspring's urine samples. A piece of bio-plastic will be placed in the diaper together with cotton balls to ensure that a sufficient amount of urine is absorbed into the cotton balls. Offspring urine will be analyzed for metabolomics.
Adult feces - Microbiome | Collected at GA34-GA36 in each pregnancy and at study visit 3, 12 and 24 months pp of 1st child
  Participants will collect a fecal spot sample at home maximum 24 hours before the planned visit.
  Will be analysed for microbiome.
Adult feces - Short chain fatty acids | Collected at GA34-GA36 in each pregnancy and at study visit 3, 12 and 24 months pp of 1st child
  Participants will collect a fecal spot sample at home maximum 24 hours before the planned visit. Will be analysed for short chain fatty acids.
Adult feces - Metabolomics | Collected at GA34-GA36 in each pregnancy and at study visit 3, 12 and 24 months pp of 1st child
  Participants will collect a fecal spot sample at home maximum 24 hours before the planned visit.
  Will be analysed for metabolomics
Adult feces - Proteomics | Collected at GA34-GA36 in each pregnancy and at study visit 3, 12 and 24 months pp of 1st child
  Participants will collect a fecal spot sample at home maximum 24 hours before the planned visit.
  Will be analysed for proteomics.
Adult feces - Inflammation markers | Collected at GA34-GA36 in each pregnancy and at study visit 3, 12 and 24 months pp of 1st child
  Participants will collect a fecal spot sample at home maximum 24 hours before the planned visit.
  Will be analysed for inflammation markers.
Adult feces - pH | Collected at GA34-GA36 in each pregnancy and at study visit 3, 12 and 24 months pp of 1st child
  Participants will collect a fecal spot sample at home maximum 24 hours before the planned visit.
  Will be assessed for pH.
Adult feces - consistency | Collected at GA34-GA36 in each pregnancy and at study visit 3, 12 and 24 months pp of 1st child
  Whenever a fecal sample is collected stool consistency of the collected sample will be collected with a questionnaire.
Adult feces - frequency | Collected at GA34-GA36 in each pregnancy and at study visit 3, 12 and 24 months pp of 1st child
  Whenever a fecal sample is collected an estimate of stool frequency during the last week will be collected with a questionnaire.
Adult feces - gastrointestinal symptoms | Collected at GA34-GA36 in each pregnancy and at study visit 3, 12 and 24 months pp of 1st child
  Whenever a fecal sample is collected gastrointestinal symptoms during the last week will be collected with a questionnaire.
Adult urine | Collected at GA34-GA36 in each pregnancy and at study visit 3, 12 and 24 months pp of 1st child
  Participants will collect a urine spot sample at the study site. Adult urine will be analyzed for metabolomics.
Offspring nutritional milestones | Collected at 12 and 18 months after offspring birth
  Parents will be instructed to register the age of the offspring when it reaches the World Health Organization (WHO) nutritional milestones (age when the offspring was introduced to specific food items)
Offspring development, WHO milestones | Collected at 12 and 18 months after offspring birth
  Parents will be instructed to register the age of the offspring when it reaches the World Health Organization (WHO) developmental milestones (age when the offspring can sit, stands in crawl-position, stands with support, stand alone, walk with support, walk alone)
Adult physical activity | Collected at study visit 3, 12 and 24 months pp of 1st child
  Physical activity and sleep will be assessed by an accelerometer and the females and males will wear the accelerometer for 7 days and 8 nights. The participants will be asked to keep a physical activity and sleep log for when they wake up and when they try to sleep
Adult physical activity - Physical Activity Questionnaire (IPAQ) | Collected at GA34-GA36 in each pregnancy, study visit at 3, 12 and 24 months pp of 1st child and 3 months pp visit after 2nd child
  Physical activity will be assessed by the International Physical Activity Questionnaire (IPAQ), in which time spent on strenuous and moderate activity and walks will be collected. The answers will be collected electronic via RedCap.
Adult background quistionnaire, ethnicity, | Collected after screening in GA34-GA36 of 1st child
  All information will be collected electronic in RedCap.
Adult background quistionnaire, education | Collected after screening in GA34-GA36 of 1st child
  All information will be collected electronic in RedCap.
Adult background quistionnaire, parity | Collected after screening in GA34-GA36 of 1st child
  All information will be collected electronic in RedCap.
Adult background quistionnaire, pre-pregnancy weight | Collected after screening in GA34-GA36 of 1st child
  Pre-pregnancy weight, ethnicity, education and parity. All information will be collected electronic in RedCap.
Adult background quistionnaire, demographic information | Collected after screening in GA34-GA36 of 1st child
  All information will be collected electronic in RedCap.
Adult wellbeing - Depression, Major depression questionnaire (ICD-10) | Collected at GA34-GA36 in each pregnancy, study visit at 3, 12 and 24 months pp of 1st child and 3 months pp visit after 2nd child
  Depression will be assessed by Major depression questionnaire (ICD-10). Mild depression: A score of 4 or 5 in two of the first three items. Plus a score of at least 3 on two or three of the last seven items.
  Moderate depression: A score of 4 or 5 in two or three of the first three items. Plus a score of at least 3 on four of the last seven items.
  Severe depression: A score of 4 or 5 in all of the first three items. Plus a score of at least 3 on five or more of the last seven items.
  Major depression: The number of items is reduced to nine, as Item 4 is part of Item 5. Include whichever of the two items has the highest score (item 4 or 5).
  A score on at least five items is required, to be scored as follows: the score on the first three items must be at least 4, and on the other items at least 3. Either Item 1 or 2 must have a score of 4 or 5.
Adult wellbeing - Quality of life, Short form-36 (SF-36) | Collected at GA34-GA36 in each pregnancy, study visit at 3, 12 and 24 months pp of 1st child and 3 months pp visit after 2nd child
  Quality of life will be assessed by the validated tool, Short form-36 (SF-36). The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Adult wellbeing - Stress, Perceived Stress Scale | Collected at GA34-GA36 in each pregnancy, study visit at 3, 12 and 24 months pp of 1st child and 3 months pp visit after 2nd child
  Stress will be assessed by validated tool, Perceived Stress Scale.Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress
Adult sleep | Collected at GA34-GA36 in each pregnancy, study visit at 3, 12 and 24 months pp of 1st child and 3 months pp visit after 2nd child
  Sleep will be assessed by the validated tool, Pittsburgh sleep quality index questionnaire (PSQI). In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Adult dietary intake, 24-h recall | Collected at GA34-GA36 in each pregnancy, at visit 3, 12 and 24 months pp of the 1st child and 3 months visit after 2nd child. Further collected at 6, 18, 30 and 36 months pp and in GA12 and GA20 of 2nd pregnancy in intervention group
  A 24 hour dietary recall is performed by a trained dietitian. Dietary recall will be registered and intake calculated using the food data program 'VITAKOST' (www.vitakost.dk).
Adult dietary intake, FFQ | Collected at GA34-GA36 in each pregnancy, at study visit 3, 12 and 24 months pp of the 1st child and 3 month follow up vist after 2nd child
  Couples will be asked to perform an electronic Food Frequency Questionnaire (FFQ). Information on frequence intake of various food groups during the last month will be collected.
Offspring dietary intake | Collected within the first week of birth and 3, 12 and 18 months after birth off each offspring
  We will collect information on offspring dietary intake including breast feeding, use of formula and type as well as use of antibiotics. The intake frequency of different foods will be collected throughout a children questionnaire.
Breast milk - nutrients biomarkers | Collected within the first week of birth and 3 months pp after each birth
  Participants will collect breast milk within the first week following birth, at 1 and 3 months pp after each birth. Participants will receive written instructions in milk collection at home. First drops will not be collected, hereafter manually expressed milk will be obtained in a sterile container. Obtained around midday and minimum two hours after last breastfeeding. Breast milk will be analyzed for nutrients biomarkers.
Breast milk - Hormonal and inflammatory markers | Collected within the first week of birth and 3 months pp after each birth
  Participants will collect breast milk within the first week following birth, at 1 and 3 months pp after each birth. Participants will receive written instructions in milk collection at home. First drops will not be collected, hereafter manually expressed milk will be obtained in a sterile container. Obtained around midday and minimum two hours after last breastfeeding. Breast milk will be analyzed for hormonal and inflammatory markers
Breast milk - Metabolomics | Collected within the first week of birth and 3 months pp after each birth
  Participants will collect breast milk within the first week following birth, at 1 and 3 months pp after each birth. Participants will receive written instructions in milk collection at home. First drops will not be collected, hereafter manually expressed milk will be obtained in a sterile container. Obtained around midday and minimum two hours after last breastfeeding. Breast milk will be analyzed for metabolomics
Breast milk - Proteomics | Collected within the first week of birth and 3 months pp after each birth
  Participants will collect breast milk within the first week following birth, at 1 and 3 months pp after each birth. Participants will receive written instructions in milk collection at home. First drops will not be collected, hereafter manually expressed milk will be obtained in a sterile container. Obtained around midday and minimum two hours after last breastfeeding. Breast milk will be analyzed for proteomics.
Breast milk - Short chain fatty acids and related metabolites | Collected within the first week of birth and 3 months pp after each birth
  Participants will collect breast milk within the first week following birth, at 1 and 3 months pp after each birth. Participants will receive written instructions in milk collection at home. First drops will not be collected, hereafter manually expressed milk will be obtained in a sterile container. Obtained around midday and minimum two hours after last breastfeeding. Breast milk will be analyzed for short chain fatty acids and related metabolites
Adult participation - dietitian guidance | Every 1-2 month from 3 months pp of 1st child to birth of 2nd child
  It will be recorded how many times of individual and group dietitian guidance the participant attends
Adult participation - physical session and power walk | Every 2nd week from 3 months pp of 1st child to birth of 2nd child
  It will be recorded how many times the participant participates in physical activity sessions and how much the person have power walked

CONTACTS AND LOCATIONS:
Overall Officials: Ulla K Opstrup, Assoc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasmussen L, Knorr S, Antoniussen CS, Bruun JM, Ovesen PG, Fuglsang J, Kampmann U. The Impact of Lifestyle, Diet and Physical Activity on Epigenetic Changes in the Offspring-A Systematic Review. Nutrients. 2021 Aug 17;13(8):2821. doi: 10.3390/nu13082821. PMID 34444981